CLINICAL TRIAL: NCT04390568
Title: An Open-label Phase I Trial to Assess Pharmacokinetics and Safety of Single Subcutaneous Doses and Single Intravenous Doses of BI 655130 in Healthy Chinese Male and Female Subjects (Single Doses, Open-label Study in Parallel-group Design).
Brief Title: A Trial in Healthy Chinese Volunteers to Test How Different Doses of BI 655130 Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0043
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Spesolimap (BI 655130) - 450 milligram (mg) - intravenous (IV) (Experimental): A single dose of 450 mg Spesolimap was administered as solution for infusion intravenously over 90 minutes (mins) after an overnight fast.
  Interventions: Drug: Spesolimap
- Spesolimap - 900 mg - IV (Experimental): A single dose of 900 mg Spesolimap was administered as solution for infusion intravenously over 90 mins after an overnight fast.
  Interventions: Drug: Spesolimap
- Spesolimap - 1200 mg - IV (Experimental): A single dose of 1200 mg Spesolimap was administered as solution for infusion intravenously over 90 mins after an overnight fast.
  Interventions: Drug: Spesolimap
- Spesolimap - 300 mg - subcutaneous (SC) (Experimental): A single dose of 300 mg Spesolimap was administered as solution for injection subcutaneously in the abdominal region within 60 seconds (s) after an overnight fast.
  Interventions: Drug: Spesolimap
- Spesolimap - 600 mg - SC (Experimental): A single dose of 600 mg Spesolimap was administered as solution for injection subcutaneously in the abdominal region within 60 s after an overnight fast.
  Interventions: Drug: Spesolimap

INTERVENTIONS:
Drug: Spesolimap — Spesolimap
  Other Names: BI 655130

SUMMARY:
The primary objective of this trial is to investigate pharmacokinetics, including dose proportionality, following single intravenous and subcutaneous doses of spesolimab in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects (at least three subjects for each gender within each dose group) according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR), body temperature), 12-lead ECG, and clinical laboratory tests.
* Chinese ethnicity, according to the following criteria: Ethnic Chinese, born in China and have 4 ethnic grandparents who were all born in China
* Age of 18 to 45 years (inclusive)
* Body weight ≥50 kg for male and ≥45 kg for female with body mass index (BMI) range ≥19 and < 26 kg/m2 at visit 1
* Signed and dated written informed consent prior to admission to the trial, in accordance with GCP and local legislation
* Female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 16 weeks after trial completion [c03320877-06]:

  * Women of childbearing potential (WOCBP)1 must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the subject information
  * A vasectomised sexual partner (vasectomy at least one year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least one year of spontaneous amenorrhoea (in questionable cases a blood sample with simultaneous levels of follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 mg/L is confirmatory)

Exclusion Criteria:

* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to treatment or planned within 12 months after screening, e.g. hip replacement
* Any finding in the medical examination (including BP, PR, RR, Body temperature or 12-lead ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic BP outside the range of 90 to 140 mmHg, diastolic BP outside the range of 50 to 90 mmHg, or PR outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including active and latent tuberculosis, human immunodeficiency virus (HIV) or viral hepatitis; QuantiFERON tuberculosis (TB) test will be performed at screening Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Cao G, Yang H, Wang J, Ishida M, Thoma C, Haeufel T, Bossert S, Zhang J. Pharmacokinetics and Safety of Spesolimab in Healthy Chinese Subjects: An Open-Label, Phase I Study. Adv Ther. 2024 Sep;41(9):3557-3568. doi: 10.1007/s12325-024-02940-8. Epub 2024 Jul 22. PMID 39039387
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label parallel-group design for intravenous (IV) and subcutaneous (SC) single-dose administration of Spesolimap (BI 655130) in healthy Chinese male and female subjects. Three cohorts were dosed consecutively in ascending order within the IV and two cohorts within the SC dose groups.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC
Started | 10 | 10 | 10 | 10 | 10
Treated | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The treatment assignment was determined based on the (first) treatment the subjects received. The treated set was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (5.8) | 31.0 (7.8) | 34.6 (5.5) | 31.5 (6.5) | 30.5 (6.9) | 31.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 4 | 20
  Male | 6 | 6 | 6 | 6 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 10 | 10 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 10 | 10 | 10 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Spesolimap in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of Spesolimap in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
  The time frames differed slightly between intravenous (IV) and subcutaneous (SC) administration. The prefix 'IV' indicates when IV was measured only. The prefix 'SC' indicates when SC was measured only. No prefix means that measurement time points were identical for IV and SC administration.
Time Frame: Within 3 hours (h) before drug administration and SC: 30 minutes (min), IV: 1h 30 min, 2h, 3h, 4h, 8h, 12h, 24h, 48h, 72h, 96h, 120h, 144h, 168h, 336h, 504h, 672h, 840h, 1008h, 1344h, 1680h, 2184h, 2856h, 3528h, 4200h after drug administration.
Population: PK parameter analysis set (PKS): This set included all participants in the treated (TS) who provided at least one primary pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. PK data from replaced participants was expected to be not evaluable and thus replaced participants were not part of the PKS. One participant (900 mg IV group) missed the last measurement time point and was removed from the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day times microgram per milliliter
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10
Day times microgram per milliliter | 3380 (17.5) | 6960 (19.2) | 10300 (21.1) | 1580 (22.2) | 3260 (34.1)
Statistical Analysis 1: Comparison: Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) vs Spesolimap - 900 mg - IV vs Spesolimap - 1200 mg - IV; No statistical hypotheses tests were planned for this trial; Test type: Other — The basic model used for the investigation of dose proportionality was a power model (regression model applied to log-transformed data) that described the functional relationship between the dose and the area under the concentration-time curve of Spesolimap in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) of the intravenous dose groups; Slope = 1.123, 90% CI 2-sided [0.979 to 1.268], Standard Error of Mean 0.085 — Based on the estimate for slope parameter (β), a 2-sided 90% confidence interval (CI) for the slope was computed. Standard error of the mean is actually standard error of slope

2. Primary Outcome: Maximum Measured Concentration of the Spesolimap in Plasma (Cmax)
Description: Maximum measured concentration of the Spesolimap in plasma (Cmax) The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
  Area under the concentration-time curve of Spesolimap in plasma over the time interval from 0 extrapolated to infinity (AUC0-8).
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
  The time frames differed slightly between intravenous (IV) and subcutaneous (SC) administration. The prefix 'IV' indicates when IV was measured only. The prefix 'SC' indicates when SC was measured only. No prefix means that measurement time points were identical for IV and SC administration.
Time Frame: as for outcome 1
Population: PK parameter analysis set (PKS): This set included all participants in the treated (TS) who provided at least one primary pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. PK data from replaced participants was expected to be not evaluable and thus replaced participants were not part of the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Groups:
- Spesolimap - 300 mg - Subcutaneous (SC): A single dose of 300 mg Spesolimap was administered as solution for injection in the abdominal region within 60 seconds (s) after an overnight fast.
- Spesolimap - 600 mg - SC: A single dose of 300 mg Spesolimap was administered as solution for injection in the abdominal region within 60 s after an overnight fast.
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Microgram per milliliter | 176 (12.5) | 370 (15.1) | 504 (17.3) | 32.0 (16.8) | 69.2 (35.7)
Statistical Analysis 1: Comparison: Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) vs Spesolimap - 900 mg - IV; No statistical hypotheses tests were planned for this trial; Test type: Other — The basic model used for the investigation of dose proportionality was a power model (regression model applied to log-transformed data) that described the functional relationship between the dose and the maximum measured concentration of the Spesolimap in plasma (Cmax) of the intravenous dose groups; Slope = 1.072, 90% CI 2-sided [0.961 to 1.183], Standard Error of Mean 0.065 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AE)s
Description: Number of participants with treatment-emergent AEs.
  All AEs occurring between first drug administration until 16 weeks thereafter were assigned to the randomised treatment.
Time Frame: Frome day of drug administration until 16 weeks thereafter, up to 16 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 8 | 9 | 8 | 7 | 9

4. Secondary Outcome: Number of Participants With Drug-related Adverse Events (AEs).
Description: Number of participants with drug-related AEs.
  All AEs occurring between first drug administration until 16 weeks thereafter were assigned to the randomised treatment.
Time Frame: Frome day of drug administration until 16 weeks thereafter, up to 16 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 4 | 8 | 4 | 4 | 7

ADVERSE EVENTS:
Time Frame: Adverse events: From the single drug administration till the end of the residual effect period, up to 113 days. All-Cause Mortality: From the single drug administration till the end of trial, up to 179 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The treatment assignment was determined based on the (first) treatment the subjects received. The treated set was used for safety analyses.
Arm/Group | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) | Spesolimap - 900 mg - IV | Spesolimap - 1200 mg - IV | Spesolimap - 300 mg - Subcutaneous (SC) | Spesolimap - 600 mg - SC
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 9/10 | 8/10 | 7/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) (N=10) | Spesolimap - 900 mg - IV (N=10) | Spesolimap - 1200 mg - IV (N=10) | Spesolimap - 300 mg - Subcutaneous (SC) (N=10) | Spesolimap - 600 mg - SC (N=10)
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimap (BI 655130) - 450 Milligram (mg) - Intravenous (IV) (N=10) | Spesolimap - 900 mg - IV (N=10) | Spesolimap - 1200 mg - IV (N=10) | Spesolimap - 300 mg - Subcutaneous (SC) (N=10) | Spesolimap - 600 mg - SC (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 2 | 0 | 0 | 0 | 0
Acne pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 0 | 1 | 4
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 2 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1 | 1 | 0 | 0
Eosinophil percentage increased (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 2 | 1 | 0 | 2
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 2
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1
Reticulocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Reticulocyte percentage increased (Investigations) | 0 | 1 | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 1 | 0
Urobilinogen urine increased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT04390568/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04390568/SAP_001.pdf